CLINICAL TRIAL: NCT05664009
Title: A Randomized, Triple-blind, Placebo Controlled, Parallel Clinical Trial to Investigate the Safety and Efficacy of Redsenol-1 Plus on Cancer-related Fatigue in Adults
Brief Title: The Safety and Efficacy of Redsenol-1 Plus on Cancer-related Fatigue in Adults
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Canada Royal Enoch Phytomedicine Co., Ltd. (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22EPRSZ03
Record Dates: First submitted 2022-12-08; First posted 2022-12-23 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Fatigue; Cancer, Treatment-Related
Keywords: Safety and efficacy; Cancer-related fatigue; Ginseng
MeSH Terms: conditions — Fatigue; Neoplasms, Second Primary

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Redsenol-1 Plus (Experimental): Participants will be instructed to take two (2) capsules, three (3) times a day in the morning, at noon and in the evening (before going to bed), for a total of 6 capsules a day, with food for 12 weeks. If a dose is missed participants are instructed to take the missed dose as soon as possible.
  Interventions: Dietary Supplement: Redsenol-1 Plus
- Placebo (Placebo Comparator): Participants will be instructed to take two (2) capsules, three (3) times a day in the morning, at noon and in the evening (before going to bed), for a total of 6 capsules a day, with food for 12 weeks. If a dose is missed participants are instructed to take the missed dose as soon as possible.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Redsenol-1 Plus — Two capsules of Redsenol-1 Plus will be taken three times per day for 12 weeks (84 days).
  Arms: Redsenol-1 Plus
Other: Placebo — Two capsules of Placebo will be taken three times per day for 12 weeks (84 days).
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of Redsenol-1 Plus on cancer-related fatigue (CRF) in adults. The change in the severity of CRF from baseline at week 12 will be assessed by the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) fatigue subscale, and compared between Redsenol-1 Plus and placebo groups. Additionally, the safety and tolerability of Redsenol-1 Plus, as compared to placebo, will be measured by the occurrence of and/or changes in treatment-emergent adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥18 years of age.
2. Females not of child-bearing potential, defined as those who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening

   Or,

   Females of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
3. Individuals previously diagnosed with cancer and have CRF defined as a score of ≥4 on the CRF Single-Item Scale (an 11-point scale where 0 is "no fatigue" and 10 is "as bad as it can be")
4. CRF present for at least one month prior to screening
5. Eastern Cooperative Oncology Group (ECOG) Performance Status Scale score ≤2
6. Hemoglobin level of ≥110 g/L for females and ≥129 g/L for males at screening
7. Agrees to maintain current lifestyle habits as much as possible throughout the study depending on ability to maintain the following: diet, medications, supplements, exercise, and sleep and avoid taking new supplements during the study period

9. Provided voluntary, written, informed consent to participate in the study

10. Otherwise healthy as determined by medical history and laboratory results as assessed by Qualified Investigator (QI) while taking into consideration the participant's cancer history

Exclusion Criteria:

1. Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
2. Allergy, sensitivity, or intolerance to the investigational product's or placebo's active or inactive ingredients
3. Individuals with any CNS malignancies (e.g., brain or spine) and/or estrogen-receptor positive breast cancer
4. Individuals with other primary causes of fatigue, as assessed by the QI (e.g., diagnosed non-cancer related chronic pain, insomnia/sleep disorders, depression/psychiatric disorders, unstable hypothyroidism, diabetes)
5. Individuals with unstable medical conditions as assessed by the QI
6. Individuals with current untreated/uncontrolled high blood pressure or tachycardia/heart rhythm disorders
7. Individuals with >7.5% HbA1c with treatment for high blood sugar/diabetes or individuals with ≥6.5% HbA1c without treatment
8. Significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case-by-case basis
9. History of or current diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones in participants who are symptom free for 6 months
10. Major non-cancer surgery in the past 3 months or individuals who have planned surgery during the course of the study. Participants with minor surgery will be considered on a case-by-case basis by the QI
11. Current use of prescription/OTC medications and/or supplements and food/drinks which may affect the efficacy and/ or safety of the IP (see Sections 7.3.1 and 7.3.2)
12. Alcohol or drug abuse within the last 12 months
13. Frequent (daily) and chronic cannabis users. Occasional (e.g., once per month) cannabis users may be included at the discretion of the QI and if eligible, asked to stop cannabis use for study period
14. Clinically significant abnormal laboratory results at screening as assessed by the QI
15. Participation in other clinical research studies 30 days prior to baseline, as assessed by the QI
16. Individuals who are unable to give informed consent
17. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant
18. Individuals who are on active cancer treatment (e.g., radiation, chemotherapy, immunotherapy, target therapy), have completed cancer treatment within one month of baseline, and/or are scheduled to receive further treatment during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The change in the severity of cancer-related fatigue from baseline to week 12. | baseline and 84 days
  The change in the severity of cancer-related fatigue from baseline to week 12 as assessed by the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) fatigue subscale will be compared between Redsenol-1 Plus and placebo.

SECONDARY OUTCOMES:
The difference in change of severity of cancer-related fatigue from baseline to weeks 4 and 8. | baseline, 28 days, 56 days
  The difference in change of severity of cancer-related fatigue from baseline to weeks 4 and 8 as assessed by the FACIT-F fatigue subscale will be compared between Redsenol-1 Plus and placebo.
The difference in change of cancer-related quality of life (QoL) from baseline at weeks 4, 8 and 12. | baseline, 28 days, 56 days, 84 days
  The difference in change of cancer-related quality of life (QoL) from baseline at weeks 4, 8 and 12 between Redsenol-1 Plus compared to placebo as assessed by the FACIT-F total score.
The difference in change of cancer-related quality of life (QoL) from baseline at weeks 4, 8 and 12. | baseline, 28 days, 56 days, 84 days
  The difference in change of cancer-related quality of life (QoL) from baseline at weeks 4, 8 and 12 between Redsenol-1 Plus compared to placebo as assessed by the FACIT-F physical well-being (PWB) sub-scale.
The difference in change of cancer-related quality of life (QoL) from baseline at weeks 4, 8 and 12. | baseline, 28 days, 56 days, 84 days
  The difference in change of cancer-related quality of life (QoL) from baseline at weeks 4, 8 and 12 between Redsenol-1 Plus compared to placebo as assessed by the social well-being (SWB) sub-scale.
The difference in change of cancer-related quality of life (QoL) from baseline at weeks 4, 8 and 12. | baseline, 28 days, 56 days, 84 days
  The difference in change of cancer-related quality of life (QoL) from baseline at weeks 4, 8 and 12 between Redsenol-1 Plus compared to placebo as assessed by the emotional well-being (EWB) sub-scale.
The difference in change of cancer-related quality of life (QoL) from baseline at weeks 4, 8 and 12. | baseline, 28 days, 56 days, 84 days
  The difference in change of cancer-related quality of life (QoL) from baseline at weeks 4, 8 and 12 between Redsenol-1 Plus compared to placebo as assessed by the functional well-being (FWB) sub-scale.
The difference in the proportion of participants who have a clinically important change in severity of cancer-related fatigue from baseline to 4 weeks, 8 weeks, and 12 weeks. | baseline, 28 days, 56 days, 84 days
  The difference in the proportion of participants who have a clinically important change in severity of cancer-related fatigue as assessed by the FACIT-F fatigue subscales from baseline to 4 weeks, 8 weeks, and 12 weeks between Redsenol-1 Plus compared to placebo.
The difference in performance status from baseline to weeks 4, 8, and 12. | baseline, 28 days, 56 days, 84 days
  The difference in performance status as assessed by the Eastern Cooperative Oncology Group (ECOG) tool from baseline to weeks 4, 8, and 12 between Redsenol-1 Plus compared to placebo.
The difference in mood from baseline to weeks 4, 8, and 12. | baseline, 28 days, 56 days, 84 days
  The difference in mood as assessed by the Profile of Mood States (POMS) questionnaire from baseline to weeks 4, 8, and 12 between Redsenol-1 Plus compared to placebo.
Incidence of pre-emergent and post-emergent adverse events following supplementation with Redsenol-1 Plus or placebo for 12 weeks. | 84 days
  Incidence of pre-emergent and post-emergent adverse events following supplementation with Redsenol-1 Plus or placebo for 12 weeks will be collected at screening and baseline and will be compared to post-emergent AEs to enable identification of AEs that may be potentially related to the investigational product.
Blood pressure at baseline and following supplementation with Redsenol-1 Plus or placebo for 4 weeks, 8 weeks, and 12 weeks. | baseline, 4 weeks, 8 weeks, 12 weeks
  Blood pressure at baseline and following supplementation with Redsenol-1 Plus or placebo for 4 weeks, 8 weeks, and 12 weeks. Blood pressure will be determined from 3 measurements obtained at least 1 minute apart. One arm will be chosen and used consistently throughout the study. Blood pressure will be checked in both arms at the first examination.
Heart rate at baseline and following supplementation with Redsenol-1 Plus or placebo for 4 weeks, 8 weeks, and 12 weeks. | baseline, 4 weeks, 8 weeks, 12 weeks
  Heart rate at baseline and following supplementation with Redsenol-1 Plus or placebo will be will be determined from 3 measurements obtained at least 1 minute apart. One arm will be chosen and used consistently throughout the study. Blood pressure will be checked in both arms at the first examination.
Aspartate aminotransferase (AST) measurement following supplementation with Redsenol-1 Plus or placebo for 12 weeks. | 84 days
  Aspartate aminotransferase (AST) will be measured in blood from study participants at 12 weeks.
Alanine aminotransferase (ALT) measurement following supplementation with Redsenol-1 Plus or placebo for 12 weeks. | 84 days
  Alanine aminotransferase (ALT) will be measured in blood from study participants at 12 weeks.
Alkaline phosphatase (ALP) measurement following supplementation with Redsenol-1 Plus or placebo for 12 weeks. | 84 days
  Alkaline phosphatase (ALP) will be measured in blood from study participants at 12 weeks.
Bilirubin measurement following supplementation with Redsenol-1 Plus or placebo for 12 weeks. | 84 days
  Total bilirubin will be measured in blood from study participants at 12 weeks.
Creatinine measurement following supplementation with Redsenol-1 Plus or placebo for 12 weeks. | 84 days
  Creatinine will be measured in blood from study participants at 12 weeks.
Measurement of electrolytes (Na, K ,Cl) following supplementation with Redsenol-1 Plus or placebo for 12 weeks. | 84 days
  Electrolytes will be measured in blood from study participants at 12 weeks.
Measurement of glucose following supplementation with Redsenol-1 Plus or placebo for 12 weeks. | 84 days
  Glucose will be measured in blood from study participants at 12 weeks.
Estimated glomerular filtration rate (eGFR) measurement following supplementation with Redsenol-1 Plus or placebo for 12 weeks. | 84 days
  Estimated glomerular filtration rate (eGFR) will be measured in blood from study participants at 12 weeks.
White blood cell count measurements following supplementation with Redsenol-1 Plus or placebo for 12 weeks. | 84 days
  White blood cell count with differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils) will be measured in blood from study participants at 12 weeks.
Red blood cell count measurements following supplementation with Redsenol-1 Plus or placebo for 12 weeks. | 84 days
  Red blood cell count will be measured in blood from study participants at 12 weeks.
Hemoglobin measurement following supplementation with Redsenol-1 Plus or placebo for 12 weeks. | 84 days
  Hemoglobin will be measured in blood from study participants at 12 weeks.
Hematocrit measurement following supplementation with Redsenol-1 Plus or placebo for 12 weeks. | 84 days
  Hematocrit will be measured in blood from study participants at 12 weeks.
Platelet count measurement following supplementation with Redsenol-1 Plus or placebo for 12 weeks. | 84 days
  Platelet count will be measured in blood from study participants at 12 weeks.
Mean corpuscular volume measurement following supplementation with Redsenol-1 Plus or placebo for 12 weeks. | 84 days
  Mean corpuscular volume will be measured in blood from study participants at 12 weeks.
Mean corpuscular hemoglobin measurement following supplementation with Redsenol-1 Plus or placebo for 12 weeks. | 84 days
  Mean corpuscular hemoglobin will be measured in blood from study participants at 12 weeks.
Mean corpuscular hemoglobin concentration measurement following supplementation with Redsenol-1 Plus or placebo for 12 weeks. | 84 days
  Mean corpuscular hemoglobin concentration will be measured in blood from study participants at 12 weeks.
Red blood cell distribution width measurement following supplementation with Redsenol-1 Plus or placebo for 12 weeks. | 84 days
  Red blood cell distribution will be measured in blood from study participants at 12 weeks.
Immature granulocyte measurement following supplementation with Redsenol-1 Plus or placebo for 12 weeks. | 84 days
  Immature granulocytes will be measured in blood from study participants at 12 weeks.
Nucleated red blood cell measurement following supplementation with Redsenol-1 Plus or placebo for 12 weeks. | 84 days
  Nucleated red blood cells will be measured in blood from study participants at 12 weeks.
Incidence of adverse events during the follow-up period (weeks 12-16). | 112 days
  Incidence of adverse events during the 4-week follow-up period (weeks 12-16).

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No